CLINICAL TRIAL: NCT02581878
Title: An Open-label Phase I, Dose-escalation Study to Evaluate the Safety, Tolerability, Maximum Tolerated Dose, Biodistribution, Radiation Dosimetry and Pharmacokinetics of BAY1862864 Injection in Subjects With Relapsed or Refractory CD22-positive Non-Hodgkin's Lymphoma
Brief Title: Safety and Tolerability of BAY1862864 Injection in Subjects With Relapsed or Refractory CD22-positive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17845; 2014-004140-36 (EudraCT Number)
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Thorium-227; BAY1862864 Injection; Safety; Pharmacokinetics; CD22; Radioimmunotherapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1a (Experimental): Cancer patients with relapsed or refractory non-Hodgkin's lymphoma will be randomized to receive an injection of study drug (BAY1862864) with a dosage of 1.5 MBq (2 mg antibody chelator conjugate [ACC]).
  Interventions: Drug: BAY1862864
- Cohort 1b (Experimental): Cancer patients with relapsed or refractory non-Hodgkin's lymphoma will be randomized to receive an injection of study drug (BAY1862864) with a dosage of 1.5 MBq (10 mg ACC).
  Interventions: Drug: BAY1862864
- Cohort 2 (Experimental): Cancer patients with relapsed or refractory non-Hodgkin's lymphoma will be randomized to receive an injection of study drug (BAY1862864) with a dosage of 3.1 MBq (10 mg ACC).
  Interventions: Drug: BAY1862864
- Cohort 3 (Experimental): Cancer patients with relapsed or refractory non-Hodgkin's lymphoma will be randomized to receive an injection of study drug (BAY1862864) with a dosage of 4.6 MBq (10 mg ACC).
  Interventions: Drug: BAY1862864
- Cohort 4 (Experimental): Cancer patients with relapsed or refractory non-Hodgkin's lymphoma will be randomized to receive an injection of study drug (BAY1862864) with a dosage of 6.1 MBq (10 mg ACC).
  Interventions: Drug: BAY1862864

INTERVENTIONS:
Drug: BAY1862864 — Radiopharmaceutical, injection: Up to four treatment cycles lasting six weeks each; in each cycle, a single treatment on Day 1. In this dose-escalation part of the study, the radioactivity dose will start at 1.5 MBq and increase in steps of 1.5 MBq, with a antibody-chelator conjugate dose of 2 or 10 mg.

SUMMARY:
To establish a recommended dose of BAY1862864 Injection and to investigate how the study drug acts in the body, on the cancer cells and how safe it is in patients with advanced non-Hodgkin's lymphoma (NHL)

DETAILED DESCRIPTION:
The study will be divided into two parts: a "dose-escalation part" to evaluate safety profile and to explore the Maximum tolerated dose (MTD) and an "expansion part" to evaluate further the safety and tumor response profile of BAY1862864 Injection at the selected dose.

ELIGIBILITY:
Inclusion Criteria:

* Subject has relapsed or refractory CD22-positive histologically confirmed NHL
* An archival paraffin-embedded tissue or fresh biopsy is available for the retrospective quantitative assessment of CD22 levels
* Bone marrow involvement of cellular marrow with lymphoma determined to be < 25%
* Subject has failed at least one prior chemo-/immunotherapy-based regimen
* Life expectancy of at least 12 weeks
* Not eligible for, or refused, or failed high-dose therapy combined with autologous stem cell rescue (HDT ASCR)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Women of childbearing potential must have negative pregnancy test within seven days before the start of treatment
* Subject was using adequate barrier birth control measures before the study and is willing to continue use of these during the entire course of the study and for the twelve months after the last administration of BAY1862864 Injection
* Adequate bone-marrow, hepatic and renal function
* Subject is capable of giving informed consent and has provided such consent in writing

Exclusion Criteria:

* Previous exposure to the study drug. Previous exposure to CD22 antibody within six months before screening. Any radio-immunotherapy within six months before screening.
* History of anaphylactic reactions to monoclonal antibody therapy. Known or suspected allergy or intolerance to any agent to be given in the course of this study.
* Anti-cancer immunotherapy and/or anti cancer chemotherapy within four weeks before the first dose of study drug
* Previous therapy with fludarabine-containing regimens within three months before screening
* Participation in any other clinical trial in which the subject received active therapy within four weeks before the first scheduled dose of study drug
* Any toxic effects (CTCAE ≥ Grade 2) of previous anti cancer therapy (incl. radiotherapy) that have not yet stabilized or significant post-treatment toxicities have been observed
* Prior definitive radiotherapy completed less than four weeks before the date scheduled for first dose of BAY1862864
* History of symptomatic metastatic brain or meningeal tumors. Presence of new or progressive brain metastases.
* History of clinically significant cardiac disease
* Clinically relevant findings in the ECG.
* Uncontrolled hypertension, defined as systolic blood pressure > 160 mmHg and / or diastolic blood pressure > 100 mmHg, despite optimum medical management
* History of arterial or venous thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, or clinically relevant pulmonary embolism within three months before the first administration of BAY1862864 (except for adequately treated catheter-related venous thrombosis occurring more than one month before start of study medication)
* Autologous bone-marrow transplant or stem-cell rescue within three months before the first administration of BAY1862864
* Organ allograft (except for corneal transplant) or allogeneic bone-marrow transplant at any time before the first administration of BAY1862864
* Positive result of hepatitis B virus (HBV-DNA) and/or human immunodeficiency virus antibody (HIV-Ab) test
* Liver cirrhosis, defined as Child-Pugh class B or C
* Any active infection of CTCAE Grade ≥2
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study
* Major surgery or significant trauma within four weeks before the first administration of BAY1862864
* Any treatment with biological response modifiers (such as, but not limited to, granulocyte colony-stimulating factor, G CSF), or any blood transfusion, within three weeks before first administration of BAY1862864
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study result
* Current pregnancy or breast-feeding
* Any condition that is unstable or could jeopardize the safety of the subject and his/her compliance with study requirements
* Close affiliation with the investigation site
* Any use by the subject of illicit drugs or other substances that may, in the opinion of the investigator or his/her designated associate(s), have a reasonable chance of contributing to toxicity or otherwise confound the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose assessed by the number of subjects with dose-limiting toxicities (DLTs) | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Skanes Universitetssjukhus, Lund, Sweden
- United Kingdom (3):
  - Southampton General Hospital, Southampton, Hampshire
  - Royal Marsden NHS Trust (Surrey), Sutton, Surrey
  - Royal Free Hospital, London

REFERENCES:
- [Derived] Linden O, Bates AT, Cunningham D, Hindorf C, Larsson E, Cleton A, Pinkert J, Huang F, Bladt F, Hennekes H, Oedegaardstuen LI, Sturm I, McNamara C. 227Th-Labeled Anti-CD22 Antibody (BAY 1862864) in Relapsed/Refractory CD22-Positive Non-Hodgkin Lymphoma: A First-in-Human, Phase I Study. Cancer Biother Radiopharm. 2021 Oct;36(8):672-681. doi: 10.1089/cbr.2020.4653. Epub 2021 Apr 21. PMID 33887152
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/